CLINICAL TRIAL: NCT05940519
Title: Short-Term Effects of Dynamic Taping on Pain, Pain Threshold, Endurance, Balance, Lumbar Joint Mobility And Functionality in Patients With Lumbar Disc Herniation
Brief Title: Short-Term Effects of Dynamic Taping in Patients With Lumbar Disc Herniation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: NAİME ULUG (Other)
Responsible Party: Sponsor-Investigator, NAİME ULUG, Assistant Professor,advisor, Atılım University
Organization: Atılım University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-59394181-604.01.02-22601
Record Dates: First submitted 2023-06-29; First posted 2023-07-11 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Lumbar Disc Herniation; Acute Pain
Keywords: lumbar disc herniation; dynamic tape; acute pain
MeSH Terms: conditions — Intervertebral Disc Displacement; Acute Pain

STUDY DESIGN:
Intervention Model Description: prospective randomized controlled study
Who Masked: Participant
Masking Description: Participant will not informed about the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dynamic tape group (Experimental): The dynamic tape group
  Interventions: Other: Dynamic taping technique; Other: Sham taping
- sham taping group (Sham Comparator): The sham tape group
  Interventions: Other: Dynamic taping technique; Other: Sham taping

INTERVENTIONS:
Other: Dynamic taping technique — The dynamic taping method as specified in the literature will be applied to the right and left lumbar paravertebral muscles in the dynamic taping group. Patients' pain will be evaluated with Numerical Rating Scale, pain threshold Jtech Commander digital algometer, lumbar muscle endurance Modified Sorenson Test, balance functional reach test, lumbar joint mobility universal goniometer and functional movement levels of patients with timed get up and go test. Evaluations will be carried out in 3 stages: before taping, 2 hours after taping and 3 days after taping. The measurements of the dynamic and sham taping applications of the 2 hours after and 3 days will be compared with the pre-taping and post taping results between two groups.
Other: Sham taping — Sham taping will be applied with a surgical patch while the patient is in a comfortable position without any technique or stretching.Evaluations will be carried out in 3 stages: before taping, 2 hours after taping and 3 days after taping. Patients' pain will be evaluated with Numerical Rating Scale, pain threshold Jtech Commander digital algometer, lumbar muscle endurance Modified Sorenson Test, balance functional reach test, lumbar joint mobility universal goniometer and functional movement levels of patients with timed get up and go test. Evaluations will be carried out in 3 stages: before taping, 2 hours after taping and 3 days after taping. The measurements of the dynamic and sham taping applications of the 2 hours after and 3 days will be compared with the pre-taping and post taping results between two groups.

SUMMARY:
Previous evidence has shown that kinesio tape application reduces pain levels and improves disability in patients with chronic low back pain due to lumbar disc herniation. However, it is not known, whether the dynamic taping can decrease back pain, improve endurance of paraspinal muscles, and improve functional capacity in patients with lumbar disk herniation. The aim of the current study is to examine the acute effects of dynamic taping on pain, pain threshold, endurance, balance, lumbar joint mobility and functionality in patients with lumbar disc herniation.

DETAILED DESCRIPTION:
The study will include 34 volunteer adult patients who have been diagnosed with lumbar disc herniation according to the physical examination and magnetic resonance imaging and have referred to the physiotherapy and rehabilitation service by a specialist physician. The patients will be divided into 2 groups as dynamic tape (n=17) and sham tape (n=17). Patients' pain will be evaluated with Numerical Rating Scale, pain threshold Jtech Commander digital algometer, lumbar muscle endurance Modified Sorenson Test, balance functional reach test, lumbar joint mobility universal goniometer and functional movement levels of patients with timed get up and go test. Evaluations will be carried out in 3 stages: before taping, 2 hours after taping and 3 days after taping. The measurements of the dynamic and sham taping applications of the 2 hours after and 3 days will be compared with the pre-taping and post taping results between two groups.

The outcomes of the study will be analyzed by appropriate statistical methods.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnose of lumbar disc herniation,
* self-reported activity pain due to lumbar disc herniation for at least the last 3 months,
* with pain severity equal to or greater than 3 on a numerical rating scale,
* patients with no skin irritation, sensitivities or allergies

Exclusion Criteria:

* Patients with spinal pathology, lumbar surgery, motor weakness, urinary or fecal incontinence due to lumbar disc herniation, cauda equina syndrome, pregnancy, neurological or rheumatological condition, dermatitis or pre-existing skin lesion over the taping area, and having dynamic taping allergies

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-07-12 (Estimated); Primary Completion 2023-08-15 (Estimated); Study Completion 2023-08-15 (Estimated)

PRIMARY OUTCOMES:
Pain severity evaluation | Up to one month
  The severity of the pain will be measured with Numerical Rating Scale. The numeric rating scale (NRS) is a pain screening tool, commonly used to assess pain severity at that moment in time using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable".
Pain threshold measurement | Up to one month
  Pain threshold will be measured Jtech Commander digital algometer

SECONDARY OUTCOMES:
The evaluation of lumbar muscle endurance | Up to one month
  Modified Sorenson Test will be used
The evaluation of balance | Up to one month
  Functional reach test will be used
Lumbar joint mobility | Up to one month
  Universal goniometer will be used
Functional movement level | Up to one month
  Timed up and go test will be used